CLINICAL TRIAL: NCT05112068
Title: Comparative Assessment of Effectiveness and Safety of Methods for Skin and Hair Care in Severe Intensive Care Unit Patients
Status: Completed | Type: Observational
Sponsor: State Budgetary Healthcare Institution, National Medical Surgical Center N.A. N.I. Pirogov, Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Other Study IDs: NMSC-01-21
Record Dates: First submitted 2021-10-13; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Pressure Ulcer
Keywords: hygienic gloves; ICU; nosocomial infections; patient skin care; pressure sores; skin lesions; critical care nursing
MeSH Terms: conditions — Pressure Ulcer; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group
  Interventions: Other: traditional skin care method
- Experimental group
  Interventions: Other: method using specialized gloves

INTERVENTIONS:
Other: traditional skin care method — Skin and hair care for critically ill patients will be carried out using traditional means: clean warm water, cotton diapers and napkins, liquid soap, 0.02% aqueous chlorhexidine solution, and regular shampoo.
  Groups: Control group
Other: method using specialized gloves — Specialized hygienic gloves soaked in a washing lotion Aqua Total Hygiene ("Cleanis", France) for skin care and Aqua Shampoo ("Cleanis", France) for hair care will be used.
  According to the manufacturer's recommendation, six hygienic gloves should be used for one skin care procedure, and two gloves should be used for hair care. The care method used in the experimental group will not require additional rinsing and drying.
  Groups: Experimental group

SUMMARY:
Skin care for seriously ill patients in the intensive care unit (ICU) is one of the key components in the prevention of serious complications that affect the treatment outcome. Bed rest, prolonged skin contact with biological secretions (urine, faeces, etc.) containing active irritating metabolic products (urea, faecal proteases, lipase, bile salts), and the use of diapers (disposable or otherwise) result in patient skin damage. Skin microbiota metabolizes urine that leads to alteration of skin pH, and promotes the propagation of opportunistic microorganisms causing infectious complications of skin and soft tissues. Additional factors, such as pressure on soft tissues, friction, or soft tissue displacement, lead to the formation of pressure sores which seriously worsens clinical results, patients' life quality, and significantly increases treatment costs. Statistics on the incidence of pressure sores in Russian medical institutions are rather scarce. It was reported that the incidence of pressure sores in hospice patients is up to 22.4%, and when assessing skin and soft tissues infections in ICU patients, the incidence of pressure sores is 28.9%.

A meta-analysis of foreign studies on the prevalence of pressure sores in ICU showed an incidence range of 7.8%-54% in studies using the methodology of the European Pressure Ulcer Advisory Panel, 6-22% in studies applying the methodology of the National Pressure Ulcer Advisory Panel, and 4.94% for a study that used the Torrance system. The probable range of the prevalence of pressure sores worldwide in intensive care facilities is from 6% to 18.5%. A recent UK randomized study found the development of new pressure sores or progression of existing ones in 15% of ICU patients with an expected stay in the ward for at least 36 hours.

Unfortunately, premorbid skin conditions that contribute to the formation of trophic disorders are largely overlooked, which results in the absence of a proper risk management system. Use of the traditional method of skin care in patients including liquid soap, napkins, and diapers can disrupt the skin barrier function and increase the risk of bedsores. This treatment method contributes to probable damage of the hydrolipid skin layer, the formation of skin microcracks, and the chemical irritation of skin, which is aggravated by frequent washing. The current trend is the use of methods that allow frequent skin washing without compromising its barrier function.

ELIGIBILITY:
Inclusion Criteria:

1. Estimated length of stay in ICU - 3 days or more.
2. Signed informed consent form.

Exclusion Criteria:

1. The presence of trophic skin changes (bedsores, maceration, intertrigo).
2. Allergy to any component of the investigated products for skin and hair care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes patients admitted to an ICU.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-09-04 (Actual); Primary Completion 2017-06-11 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
incidence rate of skin lesions | From the date of admission to the ICU until the date of discharge from ICU, assessed up to 6 months
  The incidence of skin lesions including maceration, intertrigo, excessive dryness, micro damage, and pressure ulcers at stages I-IV will be assessed daily by physical examination during the entire stay in the ICU. The incidence rate of skin trophic disorders will be estimated as a percentage after primary completion of the trial.

SECONDARY OUTCOMES:
infectious complications rate | From the date of admission to the ICU until the date of discharge from ICU, assessed up to 6 months
  The incidence of infectious complications (pneumonia, catheter-associated bloodstream infections, urinary tract infections, acute sinusitis, acute otitis) will be assessed daily during the entire stay in the ICU according to the results of diagnostic procedures (physical examination, laboratory tests and radiology procedures). The incidence rate of infectious complications will be estimated as a percentage after primary completion of the trial.
length of stay in ICU | From the date of admission to the ICU until the date of discharge from ICU, assessed up to 6 months
  Length of stay in ICU will be assessed as period of time from patient's admission to ICU to patient's transfer to another hospital unit. The mean value of this indicator measured in days will be calculated.
duration of hospitalization | From the date of admission to the hospital until the date of discharge from hospital, assessed up to 6 months
  Duration of hospitalization will be assessed as period of time from patient's admission to the hospital to patient's discharge. The mean value of this indicator measured in days will be calculated.
in-hospital mortality rate | From the date of admission to the hospital until the date of discharge from hospital, assessed up to 6 months
  in-hospital mortality rate
convenience of the investigated technique | From the date of admission to the ICU until the date of discharge from ICU, assessed up to 6 months
  Medical personnel who administered study treatment will complete a "Safety, Efficacy and Convenience of Scin Care Procedures" questionnaire daily during the entire stay of patient in the ICU. The 5-item questionnaire, which assesses the simplicity of use, degree of physical effort, possibility of use without involving additional tools, patient comfort, and nursing care time. Each characteristic (except nursing time) is rated from 1 (inadmissible) to 5 (excellent) with higher scores denoting better outcomes.
  Nursing time will be assessed in minutes and presented as median and interquartile range (Q1 - Q3).

CONTACTS AND LOCATIONS:
Locations (1):
- Pirogov National Medical and Surgical Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 6 months after completion of the study
Access Criteria: upon the request